CLINICAL TRIAL: NCT03480750
Title: Phase I Trial of Copper Chelator in Conjunction With Pegylated Liposomal Doxorubicin and Carboplatin in Patients With Platinum-resistant/-Refractory Epithelial Ovarian Cancer, Tubal Cancer and Primary Peritoneal Cancer
Brief Title: Trial of Trientine Plus Pegylated Liposomal Doxorubicin and Carboplatin in Epithelial Ovarian Cancer
Acronym: Trientine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Cheng- Yang Chou, professor, National Cheng-Kung University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-100-074
Record Dates: First submitted 2018-03-02; First posted 2018-03-29 (Actual); Results first posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Ovarian Neoplasms Malignant (Excl Germ Cell); Peritoneal Carcinoma; Fallopian Tube Cancer
Keywords: Copper chelator; Epithelial ovarian cancer; Tubal cancer; Peritoneal cancer; Trientine; Pegylated liposomal doxorubicin; Carboplatin
MeSH Terms: conditions — Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Trientine; liposomal doxorubicin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

ARMS (1):
- trientine with chemotherapy (Experimental): trientine dihydrochloride PO daily (in different dose levels) plus pegylated liposomal doxorubicin IV D1 plus carboplatin IV D1
  Interventions: Drug: trientine dihydrochloride; Drug: pegylated liposomal doxorubicin; Drug: carboplatin

INTERVENTIONS:
Drug: trientine dihydrochloride — trientine dihydrochloride 300MG/CAPSUE PO daily (in different dose levels)
  Other Names: pegylated liposomal doxorubicin; carboplatin
Drug: pegylated liposomal doxorubicin — pegylated liposomal doxorubicin 40mg/m2 IV D1
  Other Names: trientine dihydrochloride; carboplatin
Drug: carboplatin — carboplatin AUC 4 IV D1
  Other Names: trientine dihydrochloride; pegylated liposomal doxorubicin

SUMMARY:
Epithelial ovarian cancer (EOC) is the leading cause of gynecological malignancy-related deaths worldwide and is a substantial health threat to women. Many patients eventually develop chemoresistant relapsed disease and die despite surgery and combination chemotherapy. Progress in improving the survival in EOC has been slow, despite significant advances in treatment over the past 25 years. Tubal cancer and peritoneal cancer are thought to be similar in their origin, characteristics and treatment strategies. Based upon basic and animal studies, it is thought that copper chelators overcome platinum resistance. Thus, Trientine combined with carboplatin has been used to treat human cancers. The adverse effects (AEs) are acceptable in previously heavily-treated recurrent ovarian cancer patients, however, the treatment responses are limited. Therefore, here the investigators conduct a phase I trial of Trientine®, pegylated doxorubicin and carboplatin to find the dose-limited toxicities, and maximal toxicity dosage, and to explore whether the combination is applicable in epithelial ovarian, tubal and peritoneal cancers.

DETAILED DESCRIPTION:
Epithelial ovarian cancer, tubal, primary peritoneal cancers are lethal gynecologic malignances, with a 5-year survival rate below 25% for patients diagnosed with stage III-IV. Most advanced stage patients respond to cytoreductive surgery and platinum-based chemotherapy; however, >70% of women relapse, and platinum-resistant EOC is uniformly fatal. Physicians often increase the dosage of cytotoxic agents, or use single or combination second-line agents to overcome the drug resistance. Nevertheless, second-line chemotherapy sometimes may not achieve the expected cytotoxic effect and drug resistance may lead to cancer-specific death. Overcoming resistance is an important strategy for improving the therapeutic efficacy in cisplatin-containing cancer chemotherapy.

Cu homeostasis in human cells involves the inter-regulatory circuitry composed of Cu, the high-affinity Cu transporter (hCtr1) and transcription factor Sp1. Human copper transporter 1 (htr1) in humans are also involved in the import of antitumor agent cisplatin (Cp). Earlier the investigators also discovered that the magnitude of hCtr1 expression by Cu chelators depends upon the basal levels of hCtr1 expression, and that high levels of hCtr1 expression can be modulated through Cu deprivation in Cp-resistant (CpR) cells, providing a molecular basis for the development of Cu chelators as Cp resistance reversal agents in the clinical settings. D-penicillamine and Cp act synergistically to inhibit tumor growth. The investigators conduct this trial with combination agents, including LipoDox®, carboplatin and Trientine®, to develop the clinical application of copper chelator in conjunction with cytotoxic agents to conquer platinum-resistance. This trial is practical and is of perspective.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proved epithelial ovarian cancer, tubal cancer, and primary peritoneal cancer after surgical staging or debulking surgery
* The first relapse within 1 year after the completion of primary platinum-based chemotherapy (partially platinum-resistant/-sensitive) or disease progression during primary chemotherapy (platinum-refractory).
* Eastern Cooperative Oncology Group (ECOG) performance status 2 or less
* Adequate bone marrow function (absolute neutrophil count ≥ 1,500/μl, hemoglobin ≥ 9.0 g/dL and platelet count ≥ 100,000/μl)
* Serum creatinine ≤ 1.5 mg/dL or a calculated creatinine clearance of at least 50 mL/min, total serum bilirubin ≤ 5.0 mg/dL
* Alanine transaminase (ALT) or aspartate aminotransferase (AST) ≤ 5 × upper normal limit
* Patients with reproductive potential had to agree to use an effective method of birth control prior to study entry for the duration of the study participation
* If there was no available therapy that prolonged survival for at least 3 months

Exclusion Criteria:

* Patients who have metastasis to the central nervous system
* Patients who have other malignancies within 5 years prior to study entry with the exception of carcinoma in situ of the cervix uteri and non-melanoma skin cancers
* Patients who are receiving concurrent chemotherapy
* Patients who have not recovered from surgery within 4 weeks of the study;
* Patients with a clinically significant medical condition that could be aggravated by treatment or that cannot be controlled
* Patients with medical and/or psychiatric problems of sufficient severity to limit full compliance with the study or expose patients to undue risk
* Patients with known anaphylactic response or severe hypersensitivity to study drugs or their analogs
* Pregnant or lactating women
* Patients with any evidence of difficulty swallowing, intestinal obstruction or malabsorption disorder interfering with nutrition
* Patients who were unwilling or unable to provide informed consent

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female gender for gynecologic cancer (epithelial ovarian cancer, tubal cancer, and primary peritoneal cancer)
Enrollment: 18 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2019-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang YF, Kuo MT, Liu YS, Cheng YM, Wu PY, Chou CY. A Dose Escalation Study of Trientine Plus Carboplatin and Pegylated Liposomal Doxorubicin in Women With a First Relapse of Epithelial Ovarian, Tubal, and Peritoneal Cancer Within 12 Months After Platinum-Based Chemotherapy. Front Oncol. 2019 May 24;9:437. doi: 10.3389/fonc.2019.00437. eCollection 2019. PMID 31179244

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 1, 2012 and October 30, 2015, eligible patients were enrolled in a medical center, National Cheng Kung University Hospital.
Groups:
- Trientine With Chemotherapy Dose Level 1 (300mg): trientine dihydrochloride: trientine dihydrochloride 300MG/CAPSUE PO daily
  pegylated liposomal doxorubicin: pegylated liposomal doxorubicin 40mg/m2 IV D1
  carboplatin: carboplatin AUC 4 IV D1
- Trientine With Chemotherapy Dose Level 2 (600mg): trientine dihydrochloride: trientine dihydrochloride 600MG/CAPSUE PO daily
  pegylated liposomal doxorubicin: pegylated liposomal doxorubicin 40mg/m2 IV D1
  carboplatin: carboplatin AUC 4 IV D1
- Trientine With Chemotherapy Dose Level 3 (900mg): trientine dihydrochloride: trientine dihydrochloride 900MG/CAPSUE PO daily
  pegylated liposomal doxorubicin: pegylated liposomal doxorubicin 40mg/m2 IV D1
  carboplatin: carboplatin AUC 4 IV D1
- Trientine With Chemotherapy Dose Level 4 (1200mg): trientine dihydrochloride: trientine dihydrochloride 1200MG/CAPSUE PO daily
  pegylated liposomal doxorubicin: pegylated liposomal doxorubicin 40mg/m2 IV D1
  carboplatin: carboplatin AUC 4 IV D1
- Trientine With Chemotherapy Dose Level 5 (1500mg): trientine dihydrochloride: trientine dihydrochloride 1500MG/CAPSUE PO daily
  pegylated liposomal doxorubicin: pegylated liposomal doxorubicin 40mg/m2 IV D1
  carboplatin: carboplatin AUC 4 IV D1
- Trientine With Chemotherapy Dose Level 6 (1800mg): trientine dihydrochloride: trientine dihydrochloride 1800MG/CAPSUE PO daily
  pegylated liposomal doxorubicin: pegylated liposomal doxorubicin 40mg/m2 IV D1
  carboplatin: carboplatin AUC 4 IV D1
Period: Overall Study
Arm/Group | Trientine With Chemotherapy Dose Level 1 (300mg) | Trientine With Chemotherapy Dose Level 2 (600mg) | Trientine With Chemotherapy Dose Level 3 (900mg) | Trientine With Chemotherapy Dose Level 4 (1200mg) | Trientine With Chemotherapy Dose Level 5 (1500mg) | Trientine With Chemotherapy Dose Level 6 (1800mg)
Started | 3 | 4 | 3 | 3 | 3 | 2
Completed | 3 | 3 | 3 | 3 | 3 | 1
Not Completed | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — The interruption in Trientine shippment | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trientine With Chemotherapy Dose Level 1 (300mg) | Trientine With Chemotherapy Dose Level 2 (600mg) | Trientine With Chemotherapy Dose Level 3 (900mg) | Trientine With Chemotherapy Dose Level 4 (1200mg) | Trientine With Chemotherapy Dose Level 5 (1500mg) | Trientine With Chemotherapy Dose Level 6 (1800mg) | Total
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 2 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 1 | 3 | 3 | 2 | 15
  >=65 years | 1 | 0 | 2 | 0 | 0 | 0 | 3
Age, Continuous [Median (Full Range); unit: years] | 60.3 [48 to 69] | 56.3 [51 to 60] | 63.7 [47 to 74] | 50.7 [45 to 54] | 47 [44 to 49] | 56 [52 to 60] | 55.7 [44 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 3 | 3 | 2 | 18
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 3 | 3 | 3 | 2 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 3 | 4 | 3 | 3 | 3 | 2 | 18
Interval from the end of primary chemotherapy [Count of Participants; unit: Participants]
  < 6 months | 2 | 0 | 1 | 2 | 1 | 1 | 7
  6-12 months | 1 | 4 | 2 | 1 | 2 | 1 | 11
Histology [Count of Participants; unit: Participants]
  Serous adenocarcinoma | 1 | 3 | 1 | 1 | 2 | 2 | 10
  Clear cell carcinoma | 0 | 0 | 1 | 2 | 1 | 0 | 4
  Mucinous adenocarcinoma | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Mixed serous and clear cell carcinoma | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Mixed endometrioid and clear cell carcinoma | 0 | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT)
Description: (1) Grade 4 neutropenia (ANC <500/cumm^3) or thrombocytopenia ≧7 days; (2) Hematologic toxicities ≧ Grade 3, eg. febrile neutropenia <1,000/cumm^3, or platelet count <25,000/cumm^3 with hemorrhage ≧ 7 days; (3) Non-hematologic toxicities ≧ grade 3, eg. ALT or AST, ≧ 7days; other non-hematologic toxicities ≧ grade 3 (except alopecia, non-chemotherapy related nausea/vomiting); (4) Neurologic toxicities ≧ grade 2, eg. dizziness, or lethargy ≧ 3 days
Time Frame: 36 days
Population: One participant receiving 600 mg/day declined the trial drugs and did not proceed with treatment.Therefore, an additional participant was included at the same dose level.
Measure: Count of Participants; unit: Participants
Groups:
- Trientine With Chemotherapy at Dose Level 1 (300mg/d): trientine dihydrochloride PO daily plus pegylated liposomal doxorubicin IV D1 plus carboplatin IV D1
  trientine dihydrochloride: trientine dihydrochloride 300MG/CAPSUE PO daily (at 1st dose level: 300mg)
  pegylated liposomal doxorubicin: pegylated liposomal doxorubicin 40mg/m2 IV D1
  carboplatin: carboplatin AUC 4 IV D1
- Trientine With Chemotherapy at Dose Level 2 (600mg/d): rientine dihydrochloride PO daily plus pegylated liposomal doxorubicin IV D1 plus carboplatin IV D1
  trientine dihydrochloride: trientine dihydrochloride 300MG/CAPSUE PO daily (at 2nd dose level: 600mg)
  pegylated liposomal doxorubicin: pegylated liposomal doxorubicin 40mg/m2 IV D1
  carboplatin: carboplatin AUC 4 IV D1
- Trientine With Chemotherapy at Dose Level 3 (900mg/d): trientine dihydrochloride PO daily plus pegylated liposomal doxorubicin IV D1 plus carboplatin IV D1
  trientine dihydrochloride: trientine dihydrochloride 300MG/CAPSUE PO daily (at 3rd dose level: 900mg)
  pegylated liposomal doxorubicin: pegylated liposomal doxorubicin 40mg/m2 IV D1
- Trientine With Chemotherapy at Dose Level 4 (1200mg/d): trientine dihydrochloride PO daily plus pegylated liposomal doxorubicin IV D1 plus carboplatin IV D1
  trientine dihydrochloride: trientine dihydrochloride 300MG/CAPSUE PO daily (at 4th dose level: 1200mg)
  pegylated liposomal doxorubicin: pegylated liposomal doxorubicin 40mg/m2 IV D1
  carboplatin: carboplatin AUC 4 IV D1
- Trientine With Chemotherapy Dose Level 5 (1500mg/d): trientine dihydrochloride PO daily plus pegylated liposomal doxorubicin IV D1 plus carboplatin IV D1
  trientine dihydrochloride: trientine dihydrochloride 300MG/CAPSUE PO daily (at 5th dose level: 1500mg)
  pegylated liposomal doxorubicin: pegylated liposomal doxorubicin 40mg/m2 IV D1
  carboplatin: carboplatin AUC 4 IV D1
- Trientine With Chemotherapy Dose Level 6 (1800mg/d): trientine dihydrochloride PO daily plus pegylated liposomal doxorubicin IV D1 plus carboplatin IV D1
  trientine dihydrochloride: trientine dihydrochloride 300MG/CAPSUE PO daily (at 6th dose level: 1800mg)
  pegylated liposomal doxorubicin: pegylated liposomal doxorubicin 40mg/m2 IV D1
  carboplatin: carboplatin AUC 4 IV D1
Arm/Group | Trientine With Chemotherapy at Dose Level 1 (300mg/d) | Trientine With Chemotherapy at Dose Level 2 (600mg/d) | Trientine With Chemotherapy at Dose Level 3 (900mg/d) | Trientine With Chemotherapy at Dose Level 4 (1200mg/d) | Trientine With Chemotherapy Dose Level 5 (1500mg/d) | Trientine With Chemotherapy Dose Level 6 (1800mg/d)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Maximum Tolerated Dose, MTD
Description: '3+3' study design. MTD will be defined at the dose level of trientine prior to the level with DLT events ≧ 2/6 participants.
Time Frame: within 36 days after the start of Trientine
Population: as for outcome 1
Measure: Number; unit: mg
Groups:
- Trientine With Chemotherapy Dose Level 1 - 6 (300 -1800mg): trientine dihydrochloride: trientine dihydrochloride 300 - 1800MG/CAPSUE PO daily pegylated liposomal doxorubicin: pegylated liposomal doxorubicin 40mg/m2 IV D1 carboplatin: carboplatin AUC 4 IV D1
Arm/Group | Trientine With Chemotherapy Dose Level 1 - 6 (300 -1800mg)
Number analyzed (Participants) | 17
mg | NA — No DLTs or treatment-related deaths were reported, which may be due to insufficient number of participants with events to determine MTD.

3. Secondary Outcome: Maximum Plasma Concentration [Cmax] of Trientine
Description: Trientine (TETA) prior to and within 24 hrs and 7 days after trientine
Time Frame: 0, 10mins, 30mins, 60mins, 90mins, 120mins, 4h, 6h, 24h, 148h, 150h, 153h, 156h post 1st dose of trientine
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Trientine With Chemotherapy Dose Level 1 (300mg) | Trientine With Chemotherapy Dose Level 2 (600mg) | Trientine With Chemotherapy Dose Level 3 (900mg) | Trientine With Chemotherapy Dose Level 4 (1200mg) | Trientine With Chemotherapy Dose Level 5 (1500mg) | Trientine With Chemotherapy Dose Level 6 (1800mg)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2
mg/L | 1.87 [1.01 to 2.73] | 5.07 [0.83 to 9.31] | 11.54 [3.31 to 19.76] | 14.98 [8.95 to 21.01] | 13.08 [0 to 27.1] | 29.35 [0 to 29.35]

4. Secondary Outcome: Progression-free Survival
Description: Time is calculated from the diagnosis to the last follow-up date if no disease progression , or the date of disease progression after the last treatment cycle of the study drugs
Time Frame: 36 months
Population: According the protocol for this secondary outcome, data collected from participants receiving different dose levels were intended to be combined and analyzed as a single group.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Trientine With Chemotherapy: trientine dihydrochloride PO daily [through dose level 1 (300mg/day) to level 6 (1800mg/day)] plus pegylated liposomal doxorubicin IV D1 plus carboplatin IV D1
  trientine dihydrochloride: trientine dihydrochloride 300MG/CAPSUE PO daily [through dose level 1 (300mg/day) to level 6 (1800mg/day)]
  pegylated liposomal doxorubicin: pegylated liposomal doxorubicin 40mg/m2 IV D1
  carboplatin: carboplatin AUC 4 IV D1
Arm/Group | Trientine With Chemotherapy
Number analyzed (Participants) | 16
months | 4.6 [0 to 11.3]

5. Secondary Outcome: Overall Survival
Description: Time is calculated from the diagnosis to the date of the last follow-up date if no death event, or the date of death.
Time Frame: 36 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trientine With Chemotherapy
Number analyzed (Participants) | 16
months | 14.4 [0 to 34.2]

6. Secondary Outcome: Percentage of Participants With Measurable Tumor Treatment Response Assessed by RECIST Criteria 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT scan
Time Frame: 176 days
Population: Two participants who declined any of the study agents after enrollment or declined the initial chemotherapy drug after a 7-day course of trientine were deemed ineligible for this analysis. According the protocol for this secondary outcome, all participants were not described separately.
Measure: Number; unit: percentage of participants
Arm/Group | Trientine With Chemotherapy
Number analyzed (Participants) | 16
percentage of participants
  Clinical benefit rates | 43.8
  Response rates | 25.0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed up to 36 months and Serious and Other (non-serious) Adverse Events were assessed within the planned 6-month treatment duration
Description: Adverse event severity was graded according to the Common Terminology Criteria for Adverse Events, version 4.03. All participants who received at least one dose of any of the study agents were considered evaluable for safety.
Arm/Group | Trientine With Chemotherapy Dose Level 1 (300mg) | Trientine With Chemotherapy Dose Level 2 (600mg) | Trientine With Chemotherapy Dose Level 3 (900mg) | Trientine With Chemotherapy Dose Level 4 (1200mg) | Trientine With Chemotherapy Dose Level 5 (1500mg) | Trientine With Chemotherapy Dose Level 6 (1800mg)
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/3 | 3/3 | 3/3 | 3/3 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 0/3 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trientine With Chemotherapy Dose Level 1 (300mg) (N=3) | Trientine With Chemotherapy Dose Level 2 (600mg) (N=3) | Trientine With Chemotherapy Dose Level 3 (900mg) (N=3) | Trientine With Chemotherapy Dose Level 4 (1200mg) (N=3) | Trientine With Chemotherapy Dose Level 5 (1500mg) (N=3) | Trientine With Chemotherapy Dose Level 6 (1800mg) (N=2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — The only grade 4 treatment-related adverse event was thrombocytopenia, which recovered within 7 days.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trientine With Chemotherapy Dose Level 1 (300mg) (N=3) | Trientine With Chemotherapy Dose Level 2 (600mg) (N=3) | Trientine With Chemotherapy Dose Level 3 (900mg) (N=3) | Trientine With Chemotherapy Dose Level 4 (1200mg) (N=3) | Trientine With Chemotherapy Dose Level 5 (1500mg) (N=3) | Trientine With Chemotherapy Dose Level 6 (1800mg) (N=2)
Leukopenia (Investigations) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 3 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (5) | 2 (2) | 3 (6) | 3 (5) | 3 (5) | 2 (2)
Thrombocytopenia (Investigations) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (2) | 3 (3) | 3 (4) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3) | 3 (4) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (5) | 3 (5) | 3 (4) | 2 (2)
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No